CLINICAL TRIAL: NCT02598986
Title: Glycemic Index of Bread: Fiber or Minerals? This is the Question.
Brief Title: Effect of Macronutrient Supplementation on Glycemic Index of Pita Bread
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Omar Obeid, Professor, American University of Beirut Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NUT.OO.19
Record Dates: First submitted 2015-11-04; First posted 2015-11-06 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes
Keywords: glycemic index, pita bread, phosphorus, potassium, magnesium
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- white pita bread (Placebo Comparator): Pita bread made of white wheat flour
  Interventions: Dietary Supplement: Macronutrient supplementation
- Whole grain pita bread (No Intervention): no macronutrient supplementation
- Restored white pita bread (Experimental): macronutrient supplementation
  Interventions: Dietary Supplement: Macronutrient supplementation
- Fortified white pita bread (Experimental): macronutrient supplementation 2
  Interventions: Dietary Supplement: Macronutrient supplementation

INTERVENTIONS:
Dietary Supplement: Macronutrient supplementation — adding of phosphorus, potassium and magnesium
  Arms: Fortified white pita bread; Restored white pita bread; white pita bread

SUMMARY:
Glycemic index (GI) of food is known to be positively associated with the development of several diseases including type 2 diabetes, cardiovascular disease and age-related macular degeneration. Modest dietary changes from high-GI foods to low-GI foods have shown beneficial effects. These findings have been translated to recommendations for increased dietary intake of whole grains. However, the inverse relationship between whole grain consumption and risk of the different components of metabolic syndrome has not been explained by their fiber content. Trials of added cereal fiber have failed to induce a protective effect and fiber has thus been proposed to be a marker of other components of whole grains that impart health advantages. Whole wheat grains are known to be a rich source of several minerals (phosphorus, potassium and magnesium) that play a role in glucose metabolism, and are depleted during the process of refinement. Thus, it is plausible to hypothesize that the benefits of whole grains previously ascribed to their fiber content are in fact due to these minerals. The proposed research aims to restore or fortify white bread with these minerals and determine the resulting glycemic index of mineral-fortified bread. With much evidence that most people prefer the taste and color of white bread, a low GI, mineral fortified white bread has the potential to reduce the risk of Metabolic Syndrome in those who consume it.

DETAILED DESCRIPTION:
The production of white flour requires the milling of the wheat grain and extraction of a proportion of the grains. The level of 80% extraction is the most-commonly used in the production of white flour in the market and this process leads to a substantial loss of vitamins and minerals (Table 1). These vitamins and minerals are known to affect energy metabolism. For example, thiamin is known to affect carbohydrate metabolism and low thiamin intake is known to cause Beriberi. This has led to the establishment of an acceptable carbohydrate and energy: thiamin ratio (0.4mg of thiamin/1000 kcal) and many countries are fortifying their white wheat flour with thiamin to sustain an acceptable ratio. Although several minerals are known to affect energy and carbohydrate metabolism no clear ratio has been put in place yet.

Table 1: the effect of milling on mineral content of wheat flour Mineral content Wheat flour (white) Wheat flour (whole grain) Loss (%) Phosphorus (mg/100g) 108 346 69 Potassium (mg/100g) 107 408 74 Magnesium (mg/100g) 22 138 84

Specific Aim 1: Determine the acceptability of mineral fortified white bread. White flour will be supplemented with minerals to produce mineral-fortified bread. The acceptability of the bread will be tested.

White wheat flour (80% extraction) will be fortified with minerals. Potassium phosphate will be used as the source of phosphorus and potassium to fortify white flour. From previous experience, the addition of potassium phosphate to glucose solution was found to minimally affect the organoleptic properties. Unlike that of sodium phosphate that was not well tolerated by subjects due to development of unfavorable flavor (fishy flavor). At the same time, magnesium chloride will be used as the source of magnesium. Magnesium chloride is known to be highly soluble and is commonly used as a supplement or fortificant.

Locally produced white wheat flour (80% extraction) and whole grain wheat flour will be purchased and stored at the department. White and whole flour samples (n=3) will be analyzed for their content of phosphorus, magnesium and potassium according to standard procedures

Fortification:

White Bread Restoration (WB-R): A quantity of white flour will be fortified with minerals to a level that restores its content of minerals to that of whole grain wheat flour.

Based on data from the above table, white flour restoration requires the addition of:

250 mg of P/100g white flour (total P =358mg/100g) and 100 mg of Mg/100g white flour (total Mg =122mg/100g)

White Bread Fortification (WB-F): A quantity of white flour will be fortified with minerals to a level that is 100% higher than that of whole grain wheat flour.

Based on data from the above table, white flour fortification requires the addition of:

580mg of P/100g white flour (total P= 688mg/100g) 250mg of Mg/100g white flour (total Mg= 272 mg/100g)

Making of bread:

Four different types of bread will be made:

White bread (WB) White bread with mineral restoration (WB-R) White bread with mineral fortification (WB-F) Whole grain bread (WGB)

Acceptability of bread:

Bread samples (white bread and whole wheat bread controls and the 2 experimental samples) will be tested for acceptability. Panelists (n= 60) will be recruited based on their willingness to participate in the study and their consumption of Arabic bread.

Panelists will be asked to fill a questionnaire and to rate the served samples on a 9-point hedonic scale with 1 representing dislike extremely and 9 representing like extremely for overall acceptability, acceptability of appearance, texture and taste. The order of presentation of the samples will be counterbalanced.

Mineral and carbohydrate content of bread:

Phosphorus, potassium and magnesium and starch contents of the bread will be determined.

Specific Aim 2: Assess any sensory differences between the different bread treatments. The bread making step will be the same as the above. Panelists who are regular consumers of white bread will be recruited to assess any sensory differences between the white bread control and the white bread mineral supplemented experimental samples. The triangle test will be used in the difference tests. All subjects will be asked to sign human subjects consent forms and answer demographic information. Demographic information that will be requested will be: 1) age, 2) gender, 3) frequency of bread consumption, 4) type of bread typically consumed, and 5) what factors influence the panelists' bread purchase. Twenty four panelists will participate in three triangle test, comparing the white bread control vs. each of the three experimental samples in each test. In the session, subjects will be debriefed about a) the products they will consume, b) the procedures for the testing, c) instructions on how to sample the beverages, and d) how to use the score card. All samples will be presented in a random, balanced order .

Specific Aim 3: Determine the glycemic index of the mineral supplemented bread. Glycemic index of the above four different types of bread will be determined.

In this experiment, healthy subjects (n=12) will be asked to maintain their regular dietary and physical activity habits during the entire study course, avoid alcohol consumption as well as any unusual strenuous exercise 24 hours prior to the study. Exclusion criteria include: any significant medical diseases; pregnancy or lactation; regular use of medication that affects body weight; a weight loss of 3% or more in the preceding 3 months. Following a 12 hour (overnight) fast, they will be taken to the testing facility [Faculty of Agriculture and Food Sciences/Department of Nutrition or the Central research unit (CRU)/ American University Hospital] where: anthropometric measurements (height, weight) will be taken. A catheter will be inserted for blood withdrawal.

Glycemic index of food will be determined. In brief, overnight fasted subjects will be given the bread (50 g of carbohydrate) to ingest within 10-15 min and drink 250ml of water. Blood samples will be taken immediately before the meal and at 15, 30, 45, 60, 90 and 120 minutes after meal ingestion. Blood will be withdrawn by a trained practitioner and will be used for the determination of glucose.

Glucose area under the curve (AUC) will be calculated. The GI value of each food will be calculated as the mean value of : 100 x (AUC test food)/(AUC reference food) in the same subject.

In addition, mineral content of the blood will be determined and several metabolites (glucose, Tg, FFA, P), K, Mg and hormones (insulin) will be measured.

ELIGIBILITY:
Inclusion Criteria:

- Healthy subjects

Exclusion Criteria:

* any disease, pregnant and lactating

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
AUC of serum glucose | two hours